CLINICAL TRIAL: NCT00630188
Title: Shared Decision Making for Prostate Cancer Screening: a Practice-Based Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: RTI International (Other)
Responsible Party: Russell P Harris, University of North Carolina at Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TS-0845
Record Dates: First submitted 2008-02-28; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer screening; shared decision making; prostate-specific antigen; decision making; physician-patient relations
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): For Patients: Video-based decision aid on prostate cancer screening, One-on-One values clarification session with research assistant, One-on-One coaching session with research assistant to encourage good interaction with physician
  For Physicians: a one-time educational session on prostate cancer and the value of shared decision making
  Interventions: Other: You Decide
- 2 (Active Comparator): Highway Safety video
  Interventions: Other: Reducing Your Risks in the Crash

INTERVENTIONS:
Other: You Decide — For Patients: Video-based decision aid on prostate cancer screening, One-on-One values clarification session with research assistant, One-on-One coaching session with research assistant to encourage good interaction with clinician
  For Physicians: a one-time educational session on prostate cancer and the value of shared decision making
  Arms: 1
Other: Reducing Your Risks in the Crash — Publicly available video on highway safety and reducing individual risks in a crash
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether an intervention designed to help men share decisions about prostate cancer screening with their physician results in better decision making, more shared decisions, and changes in intended and actual screening rates.

DETAILED DESCRIPTION:
Background: Professional societies recommend shared decision making for prostate cancer screening, however, most effort has been directed at informed rather than shared decision making. In this study, we plan to test the effects of a shared decision making intervention on key components of shared decision making. We secondarily plan to test its effects on the presence of a shared decision, men's intention to be screened, and actual screening rates.

Methods: We plan to conduct two separate randomized controlled trials of shared decision making interventions, one in which the intervention focuses on prostate cancer screening only and one in which the intervention focuses on prostate cancer screening in the context of other men's health issues. Each trial will use the same attention control and identical implementation and measurement strategies to allow combination of data if no differences exist in the effect of the interventions. Trials will include a convenience sample of men with no prior history of prostate cancer who present to their primary care physician for routine care. Men will be randomly assigned to a shared decision making intervention (including a video and coaching session for patients and an education session for providers) or a control group, in which men will receive a video on highway safety. Data on key components of shared decision making and intent for screening will be measured at baseline, after the intervention, and after men's visit with their provider. Additionally, medical charts will be reviewed 9 months later to assess for actual screening.

ELIGIBILITY:
Inclusion Criteria:

* Ages 40-80 years
* Their physician agreed to participate in the study
* Seen in practice for at least one year

Exclusion Criteria:

* Prior history of prostate cancer
* Presenting for acute medical visit
* Non-skin cancer
* Lung disease requiring oxygen
* Renal failure requiring dialysis
* Intensive care visit in last 6 months
* Need assistance with activities of daily living

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Men's understanding that prostate cancer screening requires a decision | baseline, post intervention, post clinical visit
Men's knowledge about prostate cancer and prostate cancer screening | baseline, post intervention, post clinical visit
Men's participation in the decision about prostate cancer screening with their clinician at their preferred level | baseline, post intervention, post clinical visit

SECONDARY OUTCOMES:
The presence of a shared decision | post clinical visit
men's intent to be screened for prostate cancer | post clinical visit
Self reported screening | post visit
Actual screening by chart review | 9 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Russ Harris, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Lauren McCormack, PhD, MSPH, Principal Investigator — RTI International; David Driscoll, PhD, MSPH, Principal Investigator — RTI International
Locations (4):
- United States (4):
  - Chapel Hill North General Internal Medicine Practice, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill General Medicine Clinic, Chapel Hill, North Carolina
  - Moses Cone Internal Medicine Practice, Greensboro, North Carolina
  - Triad Internal Medicine, Greensboro, North Carolina

REFERENCES:
- [Derived] Sheridan SL, Golin C, Bunton A, Lykes JB, Schwartz B, McCormack L, Driscoll D, Bangdiwala SI, Harris RP. Shared decision making for prostate cancer screening: the results of a combined analysis of two practice-based randomized controlled trials. BMC Med Inform Decis Mak. 2012 Nov 13;12:130. doi: 10.1186/1472-6947-12-130. PMID 23148458